CLINICAL TRIAL: NCT03993210
Title: The Value of Advanced MR Imaging in Gynecological Tumors and Benign Uterine Fibroids
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Key personnel moving out
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Clare Tempany, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-056
Record Dates: First submitted 2019-05-22; First posted 2019-06-20 (Actual); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Gynecologic Tumor
Keywords: Gynecologic Tumor
MeSH Terms: conditions — Genital Neoplasms, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- GYN Cancer Cases (Experimental): * Confirmed diagnosis of primary or recurrent gynecological (GYN) malignancies.
  * Routine clinical standard of care pelvic magnetic resonance imaging (MRI) along with advanced techniques Magnetic Resonance Fingerprinting (MRF) and Q-space Trajectory Imaging (QTI) will be performed using a clinical 3T MRI scanner lasting 30-45 minutes with an additional 10-15 minutes for the advanced scans. Per protocol, patient undergoes one scan on visit day 1 and is followed for up to 4 years.
  Interventions: Device: Magnetic Resonance Fingerprinting (MRF); Device: Q-space Trajectory Imaging (QTI); Device: Magnetic Resonance Imaging Machine (MRI)
- GYN Benign Controls (Active Comparator): * Benign gynecological (GYN) fibroids.
  * Routine clinical standard of care pelvic magnetic resonance imaging (MRI) along with advanced techniques Magnetic Resonance Fingerprinting (MRF) and Q-space Trajectory Imaging (QTI) will be performed using a clinical 3T MRI scanner lasting 30-45 minutes with an additional 10-15 minutes for the advanced scans. Per protocol, patient undergoes one scan on visit day 1 and is followed for up to 4 years.
  Interventions: Device: Magnetic Resonance Fingerprinting (MRF); Device: Q-space Trajectory Imaging (QTI); Device: Magnetic Resonance Imaging Machine (MRI)

INTERVENTIONS:
Device: Magnetic Resonance Fingerprinting (MRF) — In MRF, multiple tissue properties are acquired simultaneously.
Device: Q-space Trajectory Imaging (QTI) — By using q-space trajectory encoding and a diffusion tensor distribution model, QTI improves the discrimination of diffusivity, shape, and orientation of diffusion microenvironments and therefore carries major potential for imaging the tumor microenvironment.
Device: Magnetic Resonance Imaging Machine (MRI) — MRI is routinely used in gynecologic malignancies for its ability to depict the extent of disease at diagnosis providing guidance in staging and treatment planning.

SUMMARY:
This research is being done to test new MRI methods called Magnetic Resonance Fingerprinting and Q-space Trajectory Imaging in gynecological abnormalities. The purpose of this research study is to evaluate if these new MRI methods can give additional information in characterizing gynecological tumors compared with conventional MRI.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) is a safe and painless test that uses a magnetic field and radio waves to produce detailed images of the body's organs and structures. This research is being done to test new MRI methods called Magnetic Resonance Fingerprinting (MRF) and Q-space Trajectory Imaging (QTI) in gynecological abnormalities. The purpose of this research study is to evaluate if these new MRI methods can give additional information in characterizing gynecological tumors compared with conventional MRI

In this research study, the investigators are:

* Investigating the use of MR imaging in gynecological tumors on imaging quality and comparison of tumor or fibroid structures and normal anatomy
* Investigating whether new MRI methods could help in characterizing the tumor and give information about the expected outcome

ELIGIBILITY:
Inclusion Criteria:

* Participants with suspected or histologically confirmed diagnosis of primary or recurrent gynecological cancer including uterine endometrial, cervical, vaginal, vulvar, ovarian, and smooth-muscle tumors undergoing routine clinical standard of care pelvic MRI
* Control subjects with benign fibroids undergoing routine clinical standard of care pelvic MRI
* Age ≥ 18 years
* ECOG performance status of ≤ 2, based on treating physician's discretion (Appendix A)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Contraindication to MRI identified by the MR procedure screening form, such as a pacemaker, aneurysm clip, inner ear implant, neurostimulator, or other MR non-compatible device or implant
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Adults unable to consent
* Non-english speaking subjects
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Tempany, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study closed due to PI departure.
Groups:
- Total: Total of all reporting groups
Arm/Group | GYN Cancer Cases | GYN Benign Controls | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Feasible Imaging
Description: Feasibility is determined by both A) having evaluable images in terms of quality according to radiology review and B) having a complete set of tumor metrics [MRF (T1 and T2 relaxation values) and QTI (total mean kurtosis MKT, microscopic anisotropy MKA, isotropic heterogeneity MK1, fractional anisotropy FA, microscopic fractional anisotropy µFA)]
Time Frame: Day 1
Population: No analysis was conducted because the PI left the institution. This lead to closure of the study.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: MRF T1 Relaxation Value
Description: T1 relaxation values (unit: milliseconds) will be extracted from regions-of-interest based on anatomical structures using MRF.
Time Frame: Day 1
Population: PI left the country, resulting in study closure.
Groups:
- GYN Cancer Cases: * Confirmed diagnosis of primary or recurrent gynecological (GYN) malignancies.
  * Routine clinical standard of care pelvic MRI along with advanced techniques Magnetic Resonance Fingerprinting (MRF) and Q-space Trajectory Imaging (QTI) will be performed using a clinical 3T MRI scanner lasting 30-45 minutes with an additional 10-15 minutes for the advanced scans. Per protocol, patient undergoes one scan on visit day 1 and is followed for up to 4 years.
- GYN Benign Controls: -Benign gynecological (GYN) fibroids.
  Routine clinical standard of care pelvic MRI along with advanced techniques Magnetic Resonance Fingerprinting (MRF) and Q-space Trajectory Imaging (QTI) will be performed using a clinical 3T MRI scanner lasting 30-45 minutes with an additional 10-15 minutes for the advanced scans. Per protocol, patient undergoes one scan on visit day 1 and is followed for up to 4 years.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: MRF T2 Relaxation Value
Description: T2 relaxation values (unit: milliseconds) will be extracted from regions-of-interest based on anatomical structures in using MRF.
Time Frame: Day 1
Population: PI left the country, resulting in study closure.
Groups:
- GYN Cancer Cases: * Confirmed diagnosis of primary or recurrent gynecological (GYN) malignancies.
  * Routine clinical standard of care pelvic magnetic resonance imaging (MRI) along with advanced techniques Magnetic Resonance Fingerprinting (MRF) and Q-space Trajectory Imaging (QTI) will be performed using a clinical 3T MRI scanner lasting 30-45 minutes with an additional 10-15 minutes for the advanced scans. Per protocol, patient undergoes one scan on visit day 1 and is followed for up to 4 years.
  Magnetic Resonance Fingerprinting (MRF): In MRF, multiple tissue properties are acquired simultaneously.
  Q-space Trajectory Imaging (QTI): By using q-space trajectory encoding and a diffusion tensor distribution model, QTI improves the discrimination of diffusivity, shape, and orientation of diffusion microenvironments and therefore carries major potential for imaging the tumor microenvironment.
  Magnetic Resonance Imaging Machine (MRI): MRI is routinely used in gynecologic malignancies for its ability to depict the extent of disease at diagnosis providing guidance in staging and treatment planning.
- GYN Benign Controls: * Benign gynecological (GYN) fibroids.
  * Routine clinical standard of care pelvic magnetic resonance imaging (MRI) along with advanced techniques Magnetic Resonance Fingerprinting (MRF) and Q-space Trajectory Imaging (QTI) will be performed using a clinical 3T MRI scanner lasting 30-45 minutes with an additional 10-15 minutes for the advanced scans. Per protocol, patient undergoes one scan on visit day 1 and is followed for up to 4 years.
  Magnetic Resonance Fingerprinting (MRF): In MRF, multiple tissue properties are acquired simultaneously.
  Q-space Trajectory Imaging (QTI): By using q-space trajectory encoding and a diffusion tensor distribution model, QTI improves the discrimination of diffusivity, shape, and orientation of diffusion microenvironments and therefore carries major potential for imaging the tumor microenvironment.
  Magnetic Resonance Imaging Machine (MRI): MRI is routinely used in gynecologic malignancies for its ability to depict the extent of disease at diagnosis providing guidance in staging and treatment planning.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: QTI Total Mean Kurtosis
Description: Total mean kurtosis evaluated by established methods using QTI
Time Frame: Day 1
Population: PI left the country, resulting in study closure.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: QTI Microscopic Anisotropy MKA
Description: MKa (normalized variance due to anisotropic heterogeneity, unitless) will be extracted from regions-of-interest based on anatomical structures in using advanced diffusion weighted sequences with QTI
Time Frame: Day 1
Population: PI left the country, resulting in study closure.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: QTI Isotropic Heterogeneity MK1
Description: Isotropic heterogeneity MK1 value evaluated by established methods using QTI
Time Frame: Day 1
Population: PI left the country, resulting in study closure.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: QTI Fractional Anisotropy FA
Description: Fractional anisotropy FA value evaluated by established methods using QTI
Time Frame: Day 1
Population: PI left the country, resulting in study closure.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: QTI Microscopic Fractional Anisotropy µFA
Description: Microscopic fractional anisotropy µFA value evaluated by established methods using QTI
Time Frame: Day 1
Population: PI left the country, resulting in study closure.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Median Overall Survival
Description: Time from enrollment to death or last follow-up (censored) estimated using Kaplan-Meier methods
Time Frame: Up to 4 years
Population: PI left the country, resulting in study closure.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No time frame.
Description: PI left the country, resulting in study closure. Adverse events were not assessed in this study.
Arm/Group | GYN Cancer Cases | GYN Benign Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was closed when the Principal Investigator left the country to begin work in Finland. One subject was scanned, but never analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2020-04-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03993210/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03993210/Prot_SAP_001.pdf